CLINICAL TRIAL: NCT06670170
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED CROSSOVER STUDY TO COMPARE THE SINGLE-DOSE PHARMACOKINETICS OF TWO FORMULATIONS OF PF-07976016 ADMINISTERED ORALLY TO HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn How Different Forms of the Study Medicine Called PF-07976016 Are Taken Up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C5541005; NCT06670170 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy Participants; Healthy Subjects; Human Volunteers; Normal Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Participants will receive a single dose of PF-07976016 in up to 3 study periods. In sequence 1, participants will receive formulation A followed by formulation B. There will be 7 days between each dose as a wash out period.
  Interventions: Drug: PF-07976016 Formulation A; Drug: PF-07976016 Formulation B
- Sequence 2 (Experimental): Participants will receive single doses of PF-07976016 in up to 3 study periods. In sequence 2, participants will receive formulation B followed by formulation A. There will be 7 days between each dose as a wash out period.
  Interventions: Drug: PF-07976016 Formulation A; Drug: PF-07976016 Formulation B

INTERVENTIONS:
Drug: PF-07976016 Formulation A — PF-07976016; formulation A - current/reference
Drug: PF-07976016 Formulation B — PF-07976016; Formulation B - new/test

SUMMARY:
The primary purpose of this study is to measure and compare the amount of study drug in your blood after a single dose of two formulations of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and ECG assessments.
* Willing to provide consent and follow study requirements
* Total body weight >110lbs (50kg)

Key Exclusion Criteria:

* Any condition affecting drug absorption, clinically significant laboratory values
* HIV, HepB & HepC
* Serious illness or hospitalization, or other condition, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or non-prescription drugs within a specified timeframe prior to the first dose of study intervention
* positive urine drug test at screening/admission
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening
* Use of tobacco/nicotine containing products more than the equivalent of 5 cigarettes/day or 2 chews of tobacco/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve - infinity - AUCinf (as data permit, otherwise AUClast). | Day 1 Hour 0 (pre-dose) through 168 hours post dose in each period

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events - TEAEs | From first dose (Day 1) up to 28-35 days after final dose; a total of approximately 51 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5541005